CLINICAL TRIAL: NCT04963686
Title: Simplified Assessment of Left Ventricular Systolic Function in Septic Shock Patients
Acronym: MAPSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0150
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Left Ventricular Systolic Dysfunction; Septic Shock
Keywords: Left ventricular systolic function; global longitudinal strain; Septic Shock
MeSH Terms: conditions — Ventricular Dysfunction, Left; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of left ventricular systolic function is based on the measurement of left ventricular ejection function (LVEF) by the Simpson biplane method. More recently, left ventricular global longitudinal strain (GLS) has been developed to detect abnormalities of cardiac contractility in patients with preserved myocardial contractility. However, both tools are not always easy to collect in practice. This is why other ultrasound parameters have been proposed in the literature as a substitute for LVEF and GLS such as the Doppler tissue imaging (DTI)-derived mitral annular systolic peak S-wave velocity (S'), the mitral annular plane systolic excursion (MAPSE) and the longitudinal wall fractional shortening index (LWFS).

The purpose of this project is to propose an algorithm using simple parameters (S' wave, lateral MAPSE, septal MAPSE, mean MAPSE and LWFS) to predict LVEF and GLS in order to diagnose patients with impaired systolic function and preserved ejection.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the Medical Intensive Care Department of the Amiens-Picardie University Hospital for the management of septic shock.
* Septic shock is defined by sepsis with a need for vasopressor amines to maintain a mean arterial pressure higher than or equal to 65 mmHg, and associated with hyperlactatemia (higher than 2 mmol/L).
* A transthoracic echocardiography should be performed within 72 hours of the diagnosis of septic shock.

Exclusion Criteria:

* Patient with cardiac arrhythmias,
* patients with severe mitral or aortic valve disease,
* patients with fused mitral Doppler flow,
* patients with insufficient echogenicity to allow a correct assessment of left ventricular systolic function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the Medical Intensive Care Department of the Amiens-Picardie University Hospital for the management of septic shock. Patient with a transthoracic echocardiography should be performed within 72 hours of the diagnosis of septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Concordance between LVEF and echocardiographic algorithm | 3 months
  left ventricular ejection function = LVEF The echocardiographic parameters used are: lateral S' wave; septal, lateral and mean MAPSE; and LWFS.
Concordance between GLS and echocardiographic algorithm | 3 months
  left ventricular global longitudinal strain = GLS The echocardiographic parameters used are: lateral S' wave; septal, lateral and mean MAPSE; and LWFS.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No